CLINICAL TRIAL: NCT06988878
Title: The Effect of the Flipped Learning Model on Nurses' Evidence-based Practice Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Yilidirim, MSc, BSN, PhD Student in the Department of Education in Nursing, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IstanbulUC-RN-01; Istanbul University Cerrahpasa (Other: Istanbul University Cerrahpasa)
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Evidence Based Practice; Flipped Education Model
Keywords: Education, Nursing; evidence-based practice

STUDY DESIGN:
Intervention Model Description: pre-test and post-test single group quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group that received training based on the flipped learning model (Experimental): Subjects in this group received Evidence-Based Practice Competence training based the flipped learning model once a week for six weeks.
  Interventions: Other: Evidence-based practice competence training based on the flipped learning model

INTERVENTIONS:
Other: Evidence-based practice competence training based on the flipped learning model — This training was carried out for six weeks (11 September 2024 - 16 October 2024). Once a week, participants first watched the videos uploaded by the researcher to the Edpuzzle application and participated in the offline training. Participants who had watched the videos then attended the face-to-face/traditional training. The nurse information form, the evidence-based practice knowledge test and the evidence-based practice evaluation competence questionnaire were administered to the participants before the training (4 September 2024), at the end of the training (16 October 2024) and two months after the training (18 December 2024).

SUMMARY:
The research is a quasi-experimental (intervention group) study conducted to determine the effect of 'Evidence Based Practice Competency' training based on the reverse learning model on nurses' knowledge, skills, attitudes and competencies related to evidence-based practice.

DETAILED DESCRIPTION:
Purpose: The aim of the research is to determine the effect of Evidence-Based Practice Competence training based on the reverse learning model on nurses' knowledge, skills, attitudes and competencies related to evidence-based practice.

Method: This is a quasi-experimental study with a pre-post intervention group. The research was conducted with 19 charge nurses working in a training and research hospital in Istanbul between 11 September and 18 December 2024. Data were collected using the Evidence-Based Practice Knowledge Test and the Evidence-based Practice Evaluation Competence Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Have at least a bachelor's degree in nursing

Exclusion Criteria:

* Willingness to voluntarily withdraw from the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Evidence-based Practice Evaluation Competence Questionnaire (EBP-COQ) | two months
  The scale 5-point Likert-type scale (1= Strongly Disagree, 2= Somewhat Disagree, 3= Neither Disagree nor Agree, 4= Somewhat Agree, 5= Strongly Agree) includes 25 items and three subscales (Factor 1: Knowledge, Factor 2: Skill, Factor 3: Attitudes). The statements between 1-13 form the Skills sub-dimension, the statements between 14-19 form the Attitudes sub-dimension and the statements between 20-25 form the Knowledge sub-dimension. Negative statements in the scale (items 9,10,11,15,16,18,22,24) are scored in reverse. The minimum and maximum score distributions that can be obtained from the scale are 6-30 in the Knowledge and Attitude sub-dimension, 13-65 in the Skills sub-dimension, and 25-125 overall. High scores indicate that the participant has a high level of evidence-based practice competence.
Evidence-Based Practice Knowledge Test | two months
  It consists of a total of 20 questions. Four of the questions are general information about Evidence-Based Practice, six are about asking clinical questions, one is about searching and collecting evidence, and nine are about evaluating evidence. Each question is worth five points. The lowest score that can be obtained from the knowledge test is 0, and the highest is 100. An increase in the score obtained from the test indicates that the participant has a high level of knowledge about evidence-based practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruzafa-Martinez M, Molina-Rodriguez A, Perez-Munoz V, Leal-Costa C, Ramos-Morcillo AJ. Effectiveness of the flipped classroom methodology on the learning of evidence-based practice of nursing students: Quasi-experimental design. Nurse Educ Today. 2023 Sep;128:105878. doi: 10.1016/j.nedt.2023.105878. Epub 2023 Jun 18. PMID 37352765